CLINICAL TRIAL: NCT04293731
Title: Co-administration of Smectite Gel With Live Probiotic Strains on Obesity Parameters and Insulin Resistance
Brief Title: Smectite Gel and Probiotic for Obesity and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Taras Shevchenko National University of Kyiv (Other)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO-6
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Insulin Resistance; Insulin Sensitivity; Type2 Diabetes Mellitus; Visceral Obesity
Keywords: Smectite; Probiotic; Lactobacillus; Bifidobacterium; Propionibacterium; Acetobacter; Obesity; Type2 Diabetes; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symbiter-Smectite (Active Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) per day
  Interventions: Dietary Supplement: Symbiter-Smectite
- Placebo (Placebo Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Symbiter-Smectite — Symbiter-Smectite contains biomass of alive probiotic microorganism symbiosis, colony forming units - CFU/g: Lactobacillus - 1.0х109, Bifidobacterium - 1.0х109, Lactococcus - 1.0х108, Propionibacterium - 1.0х108 and Acetobacter - 1.0х105; and smectite gel (250 mg)
  Arms: Symbiter-Smectite
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Probiotics are defined as live microorganisms that, when administered in adequate amounts, confer a health benefit on the host. Smectite is a natural silicate clay belonging to the dioctahedral smectite class formed from aluminomagnesium silicate. It is not absorbed from the gastrointestinal tract, but binds to intestinal mucous, forms multilayer structure with high plastic viscosity and powerful coating properties hence preserving integrity of the mucus, and has the ability to absorb directly bacterial toxins, bacteria, viruses and bile salts. The current study aim was to conduct placebo-controlled randomize clinical trial for the efficiency of a combination of multiprobiotics with smectite (Symbiter-Forte formulation) as an adjunction to the standard anti-diabetic therapy on IR, glycemic control parameters, β-cells functional activity, anthropometric parameters and markers of a chronic systemic inflammatory response in type 2 diabetes patients.

DETAILED DESCRIPTION:
In this single-center double-blind, placebo controlled, parallel group study, 55 type 2 diabetes patients from the Kyiv City Clinical Endocrinology Center were selected. They were randomly assigned to receive "Symbiter Smectite" or placebo for 8 weeks, administered as a sachet formulation in double-blind treatment. Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.

The "Symbiter Smectite" was supplied by Scientific and Production Company "O.D. Prolisok". It contains a biomass of alive probiotic microorganism symbiosis, colony forming units - CFU/g: Lactobacillus - 1.0х109, Bifidobacterium - 1.0х109, Lactococcus - 1.0х108, Propionibacterium - 1.0х108 and Acetobacter - 1.0х105; and smectite gel (250 mg). Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of probiotic-smectite and placebo per day. All sachets were identical with similar organoleptic characteristics (e.g., taste and appearance).

The pre-randomization period was designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study start, after inform consent signed, patients were instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants were instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent the study were instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits were provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy was compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (ages 18-75, BMI ≥25 kg/m2)
* presence of type 2 diabetes diagnosed according to criteria of the American Diabetes Association (fasting plasma glucose (FPG)≥7.0mmol/l, random plasma glucose ≥11.1mmol/l, HbA1c ≥6.5%, or glucose higher than 11.1mmol/l 2 hours after a 75-g oral glucose load);
* type 2 diabetes duration at least 6 months prior to the study;
* patient who treated with diet and exercise alone or metformin, SUs and insulin on a stabilized dose for at least 3 months before the study;
* presence of insulin resistance established as HOMA-2IR≥2.0;
* HbA1c between 6.5 and 11.0 %;
* written informed consent.

Exclusion Criteria:

* presence of type 1 diabetes;
* treatment with other than mention in inclusion criteria antidiabetic drugs (pioglitazone, GLP-1 analogues, DPP IV inhibitors etc);
* regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment;
* antibiotic use within 3 months prior to enrollment;
* allergy on probiotics or their components;
* presence of gastrointestinal diseases such as food allergy, celiac disease, non-specific ulcerative colitis;
* uncontrolled cardiovascular or respiratory disease, decompensated liver disease including ascites, encephalopathy or variceal bleeding, active malignancy, or chronic infections;
* participation in other clinical trials;
* presence of pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
HOMA-2IR | 8 weeks compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
insulin sensitivity (%S) | 8 weeks compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php

SECONDARY OUTCOMES:
HbA1c | 8 weeks compared to baseline
  HbA1c in %
fasting plasma glucose (FPG) | 8 weeks compared to baseline
  FPG in mmol/L
β-cell function (%B) | 8 weeks compared to baseline
  (%B)
C-peptide | 8 weeks compared to baseline
  C-peptide, ng/ml
weight | 8 weeks compared to baseline
  weight in kg
waist circumferences (WC) | 8 weeks compared to baseline
  WC in cm
body mass index (BMI) | 8 weeks compared to baseline
  weight in kg and height in meters will be combined to report BMI in kg/m^2
cytokines levels | 8 weeks compared to baseline
  TNF-α, IL-1β, IL-6, IL-8, INF-γ

CONTACTS AND LOCATIONS:
Overall Officials: Nazarii Kobyliak, PhD, Principal Investigator — Bogomolets National Medical University
Locations (1):
- Bogomolets National Medical University, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kobyliak N, Abenavoli L, Falalyeyeva T, Kovalchuk O, Kyriienko D, Komisarenko I. Metabolic Benefits of Probiotic Combination with Absorbent Smectite in type 2 Diabetes Patients a Randomised Controlled Trial. Rev Recent Clin Trials. 2021;16(1):109-119. doi: 10.2174/1574887115666200709141131. PMID 32646362